CLINICAL TRIAL: NCT04242147
Title: A Phase 1, Open-label, Multiple-ascending Dose Study to Investigate the Safety, Pharmacokinetics, Pharmacodynamics, and Preliminary Efficacy of KD033 (SAR445710) in Subjects With Metastatic or Locally Advanced Solid Tumors
Brief Title: A Study to Investigate the Safety, Pharmacokinetics, Pharmacodynamics, and Preliminary Efficacy of KD033 (SAR445710) in Subjects With Metastatic or Locally Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Kadmon, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TED17644; KD033-101 (Other: Kadmon); U1111-1279-2406 (Registry Identifier: ICTRP); 2022-503080-15 (Registry Identifier: CTIS); TED17644 (Other: Sanofi Identifier)
Record Dates: First submitted 2020-01-23; First posted 2020-01-27 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Bi-weekly Monotherapy Dose Escalation (Q2W) (Experimental): KD033 (SAR445710) will be administered in sequential ascending doses as a monotherapy via intravenous (IV) administration every 2 weeks (Q2W).
  Interventions: Drug: KD033 (SAR445710)
- Weekly Monotherapy Dose Escalation (Q1W) (Experimental): KD033 (SAR445710) will be administered in sequential ascending doses as a monotherapy via intravenous (IV) administration once a week (QW) for 6 weeks and then every 2 week-dosing.
  Interventions: Drug: KD033 (SAR445710)
- Dose Expansion (Experimental): KD033 (SAR445710) will be administered at recommended dose/schedule for expansion
  Interventions: Drug: KD033 (SAR445710)

INTERVENTIONS:
Drug: KD033 (SAR445710) — Pharmaceutical form: Solution for infusion Route of administration: intravenous (IV)

SUMMARY:
This is a Phase1, open-label, sequential dose-escalation and dose-expansion study of KD033 (SAR445710) in adult participants with advanced or metastatic solid tumors. The main purpose of this study is to test KD033 (SAR445710) at different dose levels to see if it is safe and well tolerated when given once every 2 weeks and when given weekly. Additional purposes of the study are to find out whether the study drug has anti-cancer effects and how the study drug is processed by the body.

DETAILED DESCRIPTION:
The foreseen treatment duration is until disease progression, unacceptable toxicity, criterion for withdrawal or for a maximum of 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed/documented advanced and/or metastatic solid tumor with at least one tumor lesion of location accessible to biopsy per clinical judgement of treating physician.
* Participants must be willing to provide a tumor biopsy at the following time points: Pre-treatment and at Cycle 4, Day 1. All other study eligibility criteria must be met before any biopsy sample is obtained.
* Measurable disease at baseline per RECIST v1.1 guidelines.
* Life expectancy of at least 3 months.
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) score ≤ 1.
* Adequate organ and bone marrow functions.
* All toxicities related to prior radiotherapy, chemotherapy, or surgical procedure must have recovered to baseline or Grade ≤ 1 based on NCI-CTCAE v5.0 except alopecia (any grade), Grade 2 peripheral neuropathy and adverse events that are clinically non-significant or stable on supportive care.
* All participants, male and female, who are not surgically sterilized or postmenopausal must agree to use 'highly effective methods of contraception' during the study and for at least 60 days after the last dose of KD033 (SAR445710).
* Women of childbearing potential must have a negative pregnancy test within 7 days prior to KD033 (SAR445710) treatment.
* Ability to understand the purpose of the study, provide signed and dated informed consent from the participant/legal representative prior to performing any protocol-related procedures and able to comply with the study procedures and any locally required authorization.

Exclusion Criteria:

* Use of immunotherapy, biological therapy, cytokine therapy < 21 days prior to the first dose of study drug.
* Use of immunomodulating agents < 21 days prior to the first dose of study drug.
* Use of chemotherapy and approved tyrosine kinase inhibitor (TKI) therapy < 14 days prior to the first dose of study drug.
* Anti PD-L1 or anti PD-1 therapy < 6 weeks prior to the first dose of study drug.
* Radiotherapy within 14 days before the start of trial treatment (prior diagnostic biopsy is permitted), with the exception of palliative radiation as described: patients assigned to radiotherapy require at least 1 additional lesion that can be safely irradiated while sparing the index lesion(s), and for which radiation at the limited, palliative doses contemplated would be considered medically appropriate; The lesion should be causing some signs or symptoms (e.g., tumor-related pain), for which radiation is indicated per the physician's standard clinical practice.
* Use of any investigational drug or have major surgery within 28 days before the start of trial treatment
* Ongoing or recent (within 2 years) evidence of significant autoimmune disease that required systemic immunosuppressive treatments.
* Systemic therapy with immunosuppressive agents including corticosteroids within 14 days before the start of trial treatment with the exception of corticosteroid replacement therapy for adrenal insufficiency
* Rapidly progressive disease which, in the opinion of Investigator, may predispose to inability to tolerate treatment or trial procedure.
* History or clinical evidence of central nervous system primary tumors or metastases including leptomeningeal metastases unless they have been previously treated, demonstrated no progression at least 1 months, are asymptomatic and have had no requirement for steroids or enzyme inducing anticonvulsants in the last 14 days before Screening - Participants with suspected brain metastases at Screening should undergo a CT/MRI of the brain prior to study entry.
* Receipt of any organ transplantation including hematopoietic cell transplantation.
* Has a paraneoplastic syndrome of autoimmune nature.
* History of interstitial lung disease or severe obstructive pulmonary disease.
* Clinically significant cardiovascular/cerebrovascular disease.
* QTc(F) interval > 450 ms for men or > 470 ms for women)
* Left ventricular ejection fraction (LVEF) < 50% as measured by an echocardiogram (ECHO).
* Active infection requiring therapy.
* Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding.
* Pregnant or breast-feeding women
* Known severe hypersensitivity reactions to monoclonal antibodies, any history of or recent (within 6 months) of anaphylaxis
* Vaccine administration within 4 weeks of investigational drug administration.
* Vaccination with live vaccines while on trial is prohibited. Administration of inactivated vaccines like inactivated influenza vaccines is allowed. COVID-19 vaccines are approved to be administered prior to KD033 (SAR445710) administration and during the treatment phase, however, it is preferred to not vaccinate during the 28-day DLT period.

Note: Other protocol-defined exclusion criteria could apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2023-03-06 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Occurrence of Dose Limiting Toxicities (DLTs) | Up to 28 days
  To evaluate the number of participants who experienced DLTs during the dose escalation phase
Treatment Emergent Adverse Events (TEAEs) and Treatment-related AEs by Severity | Up to 30 days after last treatment
  To evaluate the number of TEAEs and treatment-related AEs by severity for all dose groups/cohorts according to the National Cancer Institute Common Terminology Criteria for Adverse Events Version 5.0 (NCI CTCAE v5.0)

SECONDARY OUTCOMES:
Best Overall Response (BOR) | Through study completion, an expected average of 1 year
  To evaluate the best overall response from study treatment according to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) and Immune Response Evaluation Criteria in Solid Tumors (iRECIST) criteria per Investigator assessment
Duration Of Response (DOR) | Through study completion, an expected average of 1 year
  To evaluate the duration of response from study treatment according to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) and Immune Response Evaluation Criteria in Solid Tumors (iRECIST) criteria per Investigator assessment
Exploration of KD033 (SAR445710) Pharmacokinetic (PK) Profile - AUC | Through study completion, an expected average of 1 year
  Area under the concentration versus time curve (AUC)
Exploration of KD033 (SAR445710) Pharmacokinetic (PK) Profile - Cmax | Through study completion, an expected average of 1 year
  Maximum plasma concentration observed (Cmax)
Exploration of Anti-KD033 (SAR445710) Antibodies | Through study completion, an expected average of 1 year
  To evaluate serum titers and assessment of neutralization of anti-KD033 (SAR445710) antibodies using blood samples collected during the dose escalation and dose expansion phases

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - UCLA Hematology/Oncology, 2020 Santa Monica Boulevard, Suite 600 - Site 042, Santa Monica, California
  - Moffitt Cancer Center - Site 102, Tampa, Florida
  - Roswell Park Cancer Institute - 665 Elm St - Site 062, Buffalo, New York
  - Fox Chase Cancer Center - 333 Cottman Avenue - Site 141, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center - Hillman Cancer Center - 5150 Centre Avenue, Suite 301 - Site 132, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: TED17644 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25764&tenant=MT_SNY_9011